CLINICAL TRIAL: NCT03034239
Title: The Effect of Insect Protein on Performance and Hypertrophy During Eight Weeks of Resistance Training
Brief Title: The Effect of Insect Protein on Performance and Hypertrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Insect2017
Record Dates: First submitted 2017-01-23; First posted 2017-01-27 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-01

CONDITIONS: Protein Supplementation
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insect protein group (Experimental): Exercise + insect protein 8 weeks of 4/week progressive resistance training (2 days upper body, 2 days lower body). Insect protein supplementation (4g/kg) after each training + before sleep at training days, and once in the morning at non training days.
  Interventions: Dietary Supplement: Protein supplementation; Other: Resistance training
- Placebo group (Placebo Comparator): Exercise + isocaloric carbohydrate 8 weeks of 4/week progressive resistance training (2 days upper body, 2 days lower body). Carbohydrate supplementation (isocaloric to protein group) after each training + before sleep at training days, and once in the morning at non training days.
  Interventions: Other: Resistance training

INTERVENTIONS:
Dietary Supplement: Protein supplementation — + insect protein
  Arms: Insect protein group
Other: Resistance training — Resistance exercise

SUMMARY:
Purpose: to study the effect of insect protein on performance and hypertrophy during 8 weeks of resistance training.

Hypothesis: Insect protein supplementation enhances the effect of resistance training on muscle mass and muscle strength.

Primary outcome: Muscle hypertrophy and muscle strength

Design: Two groups of healthy young men (age: 18-30 years) with resistance training experience, but no structural resistance training performed for the last 12 months. Randomized controlled intervention study +/- insect protein (placebo group ingest isocaloric carbohydrate). Both groups perform 8 weeks of progressive resistance training (4/week) aiming to induce muscle hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young men (age: 18-30 years) with experience in resistance training
* 2 hours of physical exercise per week or more

Exclusion Criteria:

* No structural resistance training for the last 12 months
* No injuries
* No smoking
* No ingesting of protein or creating supplementations
* No use of medicine which may influence the adaptation to strength training

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Muscle hypertrophy | 8 weeks
  muscle mass measured by DXA-scan

SECONDARY OUTCOMES:
Muscle Strength | 8 weeks
  muscle strength measured by maximal isometric muscle strength, 1RM at bench press and leg press and 80% 1RM to fatigue in bech and leg press

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hansen, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark